CLINICAL TRIAL: NCT04178304
Title: Effect of Prolotherapy in Knee Osteoarthritis: Clinical and Ultrasonographic Study.
Brief Title: Effect of Prolotherapy in Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Yousra Hisham Abdel Fattah, Lecturer of Physical Medicine, Rheumatology and Rehabilitation, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0201167
Record Dates: First submitted 2019-11-21; First posted 2019-11-26 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
Keywords: primary knee osteoarthritis,; prolotherapy,; musculoskeletal ultrasound
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Prolotherapy; Glucose

STUDY DESIGN:
Intervention Model Description: Sixty knees with primary knee osteoarthritis will be included in the study, plain X-ray for the affected knee, followed by musculoskeletal ultrasound assessment will be done. The intervention: 1. a single intra-articular injection of 6 mL of 25% dextrose through infero-medial or infero-lateral approach will be done. 2. extra-articular injections will be done at major tender tendons and ligaments through 15 skin punctures using peppering technique and placing a possible total of 22.5 mL of 25% dextrose. Both intra and extra-articular injections will be done at 1, 5, 9, and 13 weeks intervals. Follow up will be done at 24 weeks after the last injection both clinically and ultrasounographicly.
Masking Description: the Assessor doing the musculoskeletal ultrasound will be masked to the radiographic grading of knee osteoarthritis, the clinical condition and the improvement following prolotgerapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- G1 patients receive prolotherapy (Experimental): Intra and extra articular dextrose 25%
  Interventions: Drug: Prolotherapy with 25% Dextrose

INTERVENTIONS:
Drug: Prolotherapy with 25% Dextrose — Intra-articular injection of 6mL of 25% dextrose Extra-articular injection at tender sites with 25% dextrose
  Other Names: 25% dextrose intra and extra-articilar injection

SUMMARY:
Patients with primary knee osteoarthritis will be included in the study, plain X-ray for the affected knee, followed by musculoskeletal ultrasound assessment will be done. The intervention: intra-articular injection and extra-articular injections of 25% dextrose. Follow up will be done at 24 weeks after the last injection both clinically and ultrasonographically .

Aim: Determine whether prolotherapy improves pain. stiffness and function of symptomatic knee osteoarthritis and determine ultrasonographic changes before and after prolotherapy.

DETAILED DESCRIPTION:
Sixty knees with primary knee osteoarthritis will be included in the study, clinical assessment will be done, then plain X-ray for the affected knee (s), followed by musculoskeletal ultrasound assessment will be done.

The intervention:

1. a single intra-articular injection of 6 mL of 25% dextrose through infero-medial or infero-lateral approach will be done.
2. extra-articular injections will be done at major tender tendons and ligaments through 15 skin punctures using peppering technique and placing a possible total of 22.5 mL of 25% dextrose.

   * Both intra and extra-articular injections will be done at 1, 5, 9, and 13 weeks intervals.

Follow up will be done at 24 weeks after the last injection both clinically and ultrasonographically .

ELIGIBILITY:
Inclusion Criteria:

* Moderate and moderate to severe primary Knee osteoarthritis (KL grade II and III)
* consent obtained

Exclusion Criteria:

* Early Knee osteoarthritis (KL grade I)
* Severe Knee osteoarthritis (KL grade IV)
* Causes of 2ry osteoarthritis: other rheumatological, metabolic and inflammatory joint diseases.
* received oral or systemic steroids 1 year prior to the procedure
* received intra-articular steroids or hyaluronic acid 1 year prior to the procedure
* BMI >45Kg/m2
* poorly controlled diabetes mellitus, on anticoagulation therapy, history of cancer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Pain, Stiffness and Physical function | 24 weeks after last injection
  whether prolotherapy improves physical function by Western Ontario and McMaster University (WOMAC) index and VAS in patients with primary knee osteoarthritis

SECONDARY OUTCOMES:
Cartilage thickness | 24 weeks after last injection
  whether an increase in cartilage thickness could be detected by the musculoskeletal ultrasound following prolotherapy
Safety and Tolerability | 24 weeks after last injection
  safety and tolerability will be assessed using patient satisfaction Likeret 5 point scale

CONTACTS AND LOCATIONS:
Overall Officials: Yousra H Abdel-Fattah, MD, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No